CLINICAL TRIAL: NCT06701201
Title: A Long-Term Follow-Up Basket Study for Participants Treated With SynKIR Chimeric Antigen Receptor (CAR) T Cell Product
Status: Enrolling by invitation | Type: Observational
Sponsor: Verismo Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: LTFU 101-00
Record Dates: First submitted 2024-11-18; First posted 2024-11-22 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Cancer
Keywords: Cancer; CAR-T; CAR-T Cells; KIR-CAR
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SynKIR-110: Participants who previously received SynKIR-110 in an interventional trial
  Interventions: Drug: SynKIR-110
- SynKIR-310: Participants who previously received SynKIR-310 in an interventional trial
  Interventions: Drug: SynKIR-310

INTERVENTIONS:
Drug: SynKIR-110 — Autologous T cells Transduced with Mesothelin KIR-CAR
  Groups: SynKIR-110
Drug: SynKIR-310 — Autologous T Cells transduced with CD19 KIR-CAR
  Groups: SynKIR-310

SUMMARY:
The primary purpose of this study is to monitor potential long-term risks associated with the administration of SynKIR CAR T cell products.

DETAILED DESCRIPTION:
This is a study for the Long Term Follow Up for all participants treated with Verismo Therapeutics' SynKIR CAR T cell products in accordance with regulatory guidance. The primary objective of this study is to monitor the long-term safety of SynKIR CAR T cell products.

No investigational product will be administered in this LTFU study. Eligible participants must have received at least 1 infusion of a SynKIR CAR T cell product under a Verismo Therapeutics parent protocol. Participants will be invited to enroll into this LTFU study after either early discontinuation from or completion of the parent protocol.

In accordance with regulatory guidelines, this study will follow participants for a period of 15 years following infusion of Verismo Therapeutics' SynKIR CAR T cell product, to monitor for delayed adverse events (AEs), detection of replication competent lentivirus (RCL), and to assess long-term efficacy and persistence of gene-modified T cells.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

1. All adult participants who have received any amount of SynKIR CAR T cell product in a study sponsored by Verismo Therapeutics.
2. Participant is willing and able to comply with the study requirements.

Exclusion Criteria:

There are no specific exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants must have received at least 1 infusion of a SynKIR CAR T cell product in a Verismo Therapeutics parent protocol.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2042-02 (Estimated); Study Completion 2042-02 (Estimated)

PRIMARY OUTCOMES:
To monitor the long-term safety of participants that have been infused with a SynKIR CAR T cell product | Up to 15 years from SynKIR CAR T cell product administration
  Frequency and severity of delayed AEs considered related to SynKIR CAR T cell product
To monitor the long-term safety of participants that have been infused with a SynKIR CAR cell product | Up to 15 years from SynKIR CAR T cell product administration
  Presence of RCL VSV-G DNA

SECONDARY OUTCOMES:
To assess the long-term clinical efficacy of SynKIR CAR T cell product | Up to 15 years from SynKIR CAR T cell product administration
  Overall survival
To assess the long-term clinical efficacy of SynKIR CAR T cell product | Up to 15 years from SynKIR CAR T cell product administration
  Progression-free survival
To assess the persistence of SynKIR-modified T cells | Up to 15 years from SynKIR CAR T cell product administration
  Presence of a SynKIR CAR DNA sequence

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Colorado Blood Cancer Institute, part of Sarah Cannon Research Institute, Denver, Colorado
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - University of Kansas Cancer Center, Westwood, Kansas
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin